CLINICAL TRIAL: NCT05855759
Title: Acellular Matrix Homologous From Human Dermis in Combination With Orthobiologic Stimuli,Subacromial Bursa and Humeral Bone Marrow Concentrate, for Augmentation of Massiverotator Cuff Tears: Therapeutic Efficacy and Improvements for the Development of a Costeffective and Ready to Use Product
Brief Title: Acellular Matrix From Human Dermis in Combination With Orthobiologic Stimuli for Augmentation of Massive Rotator Cuff Tears
Acronym: MODA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MODA
Record Dates: First submitted 2023-04-14; First posted 2023-05-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acellular Dermal Matrix (Active Comparator): Enrolled patients will be randomly assigned to the suture-bridge technique with acellular dermal matrix
  Interventions: Other: Acellular Dermal Matrix
- Acellular Dermal Matrix with autologous orthobiologics (Experimental): Enrolled patients will be randomly assigned to the suture-bridge technique with acellular dermal matrix with orthobiologics autologous: humeral bone marrow concentrate and subacromial bursa
  Interventions: Other: Acellular Dermal Matrix with autologous orthobiologics

INTERVENTIONS:
Other: Acellular Dermal Matrix — Patinets will be treated with acellular dermal matrix with standard arthroscopic technique performed as per normal clinical practice. For the tendon repair the acellular dermal matrix patch will be placed over the repaired tendon with dedicated sutures and anchors.
  Arms: Acellular Dermal Matrix
Other: Acellular Dermal Matrix with autologous orthobiologics — Patinets will be treated with acellular dermal matrix enriched with autologous humeral bone marrow concentrate and subacromial bursa with standard arthroscopic technique. Humeral bone marrow concentrate will be harvested from the proximal humeral head inthe operating room and concentrated by an automatic close system.
  Arms: Acellular Dermal Matrix with autologous orthobiologics

SUMMARY:
The use of biologic acellular matrices for the surgical augmentation of rotator cuff lesions has greatly expanded inrecent years. The study team patented a method for removing cells from human dermis (Acellular Dermal Matrix), maintaining unaltered biological and structural integrity. Acellular Dermal Matrix has been succesfully used for rotator cuff surgical repair augmentation beside in a limited number of patients. The aim of the project is to demonstrate the therapeutical efficacy of this strategy in patients affected by rotator cuff massive tears. Acellular Dermal Matrix will be also combined with autologous orthobiologics.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by large to massive lesion according to Gerber involving supraspinatus and infraspinatus tendons
* tendon retraction <=3 according to Thomazeau
* fatty degeneration <=3 according to Goutallier
* possibility to obtain tendon reduction,
* pre-operative Magnetic Resonance Imaging,
* ability to read, understand and complete outcome scores

Exclusion Criteria:

* patients affected by osteoarthritic degeneration,
* frozen shoulder,
* symptomatic acromioclavicular arthritis,
* revision surgeries,
* inability to cope with post-operative rehabilitation regimen,
* autoimmune connective tissue disease,
* current or past hematologicaldisorders,
* comorbidities affecting healing,
* active infections,
* cancers,
* pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
re-tear rate | 12 months after surgery
  Presence/absence of re-tear on magnetic resonance imaging

SECONDARY OUTCOMES:
cell yeld | baseline
  number of stromals cells contained in the humeral bone marrow concentrate
subacromial bursa | baseline
  Half of the subacromial bursal tissue wll be assessed for determining the cell yield (number of stromal cells contained for mg of tissue) and half for histological processing

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

REFERENCES:
- [Result] Rotini R, Marinelli A, Guerra E, Bettelli G, Castagna A, Fini M, Bondioli E, Busacca M. Human dermal matrix scaffold augmentation for large and massive rotator cuff repairs: preliminary clinical and MRI results at 1-year follow-up. Musculoskelet Surg. 2011 Jul;95 Suppl 1:S13-23. doi: 10.1007/s12306-011-0141-8. PMID 21691735
- [Result] Bondioli E, Fini M, Veronesi F, Giavaresi G, Tschon M, Cenacchi G, Cerasoli S, Giardino R, Melandri D. Development and evaluation of a decellularized membrane from human dermis. J Tissue Eng Regen Med. 2014 Apr;8(4):325-36. doi: 10.1002/term.1530. Epub 2012 Jun 11. PMID 22689414